CLINICAL TRIAL: NCT00004446
Title: Study of Fluoxetine in Patients With Depersonalization Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/13456; MTS-GCO-95-323
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-03

CONDITIONS: Depersonalization Disorder
Keywords: depersonalization disorder; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Depersonalization; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Fluoxetine

INTERVENTIONS:
Drug: fluoxetine

SUMMARY:
The purpose of this study is to:

1) Determine the effects of fluoxetine in the treatment of depersonalization disorder, 2) Assess the durability of treatment response in these patients, 3) Assess the improvement in psychiatric disability in these patients, and 4) Assess the effects of comorbid Axis I disorders (depression, social phobia, panic/anxiety, obsessive-compulsive disorder) and Axis II personality disorders on treatment outcome in these patients.

DETAILED DESCRIPTION:
In this trial, participants will be randomly assigned to receive either fluoxetine or placebo. Treatment will consists of two phases (acute treatment and maintenance). In the acute treatment phase, participants will receive fluoxetine or placebo daily for 12 weeks. Participants will be followed every 2 weeks. In the Maintenance phase, participants showing significant improvement after 12 weeks may continue treatment for an additional 6 months. In this phase, participants are followed every 4 weeks.

Participants who do not improve during the acute treatment phase may receive open fluoxetine, or another appropriate medication, for 3 months.

ELIGIBILITY:
Inclusioin Criteria:

* Meets DSM-IV criteria for depersonalization disorder in the last month

Exclusion Criteria:

* Prior or concurrent bio- or chemotherapy or
* Use of any of the following within 2 weeks prior to study entry: antipsychotics, anticonvulsants, stimulants, barbiturates, lithium, benzodiazepines, or antidepressants
* Use of MAO inhibitors or investigational drugs within 4 weeks prior to study entry
* History of fluoxetine use at a dose of 10 mg or more for at least 6 weeks duration
* Hematologic, hepatic, renal, cardiovascular, pulmonary, metabolic, endocrine, systemic, or gastrointestinal disease
* History of mental disorders
* Current substance abuse
* Current eating disorder
* Current clinically unstable suicidal ideation
* Unstable medical illness
* Clinically unstable
* Clinically important abnormalities in lab tests or physical exams
* History of seizure disorders or abnormal electroencephalogram
* Hypersensitivity or severe side effects to fluoxetine
* Pregnancy or breast-feeding. Women of child-bearing potential must use effective contraception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 1998-04

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Simeon, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Medical Center, NY, New York, New York, United States

REFERENCES:
- [Background] Simeon D, Guralnik O, Schmeidler J, Knutelska M. Fluoxetine therapy in depersonalisation disorder: randomised controlled trial. Br J Psychiatry. 2004 Jul;185:31-6. doi: 10.1192/bjp.185.1.31. PMID 15231553